CLINICAL TRIAL: NCT02634593
Title: The Snack Study: The Feasibility of Changing Night-time Food Choices to Improve Glucose Tolerance in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paula Chandler-Laney, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: F140825002; R03DK104010 (NIH)
Record Dates: First submitted 2015-12-10; First posted 2015-12-18 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Glucose Intolerance; Obesity
Keywords: nutrition
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control
- Low glycemin load snacks (Active Comparator): Low glycemic load snacks, consumed during specific times
  Interventions: Behavioral: Low glycemic load snacks

INTERVENTIONS:
Behavioral: Low glycemic load snacks — Intervention to replace standard night-time food and drinks with lower glycemic load options
  Arms: Low glycemin load snacks

SUMMARY:
Obesity during pregnancy increases the risk for high glucose and diabetes in the mother, and for obesity and comorbid metabolic disease in the offspring. Results of previous intervention studies designed to improve the metabolic health of obese mothers, and thereby reduce the risk to their offspring, have been modest at best. Furthermore, few studies have proved to be efficacious among low income African American women who have high risk for the transmission of obesity to future generations. The purpose of this study is to examine the feasibility of changing the types of foods and drinks that are consumed at night during late pregnancy in order to improve maternal glucose tolerance and reduce the risk for future obesity in the child.

DETAILED DESCRIPTION:
Obesity during pregnancy increases the risk for high glucose and diabetes in the mother, and for obesity and comorbid metabolic disease in the offspring. Results of previous intervention studies designed to improve the metabolic health of obese mothers, and thereby reduce the risk to their offspring, have been modest at best. Furthermore, few studies have proved to be efficacious among low income African American women who have high risk for the transmission of obesity to future generations. The purpose of this study is to examine the feasibility of changing the types of foods and drinks that are consumed at night during late pregnancy in order to improve maternal glucose tolerance and reduce the risk for future obesity in the child. We hypothesize that women who replace their usual night-time foods and drinks with lower glycemic load options will have more stable night-time glucose and lower glucose following an oral glucose load. This intervention will be assessed in a cohort of African American women of low income, who were obese at their first prenatal care visit.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* Healthy, singleton pregnancy
* ≤ 28 weeks' gestation at enrollment
* BMI of 30.0 - 45.9 kg/m2 at first prenatal visit
* Reports regular food consumption after 8pm at night that is not attributable to work schedule or other constraints.

Exclusion Criteria:

* pre-gestation or gestational diabetes
* current smoker
* presence of any medical condition or the use of any medication known to affect fetal growth
* previous delivery of a small-for-gestational age infant (<10th percentile)
* previous delivery of a pre-term infant (<36.0 weeks' gestation)
* inability to communicate in both verbal and written English
* unwilling or unable to consume study-provided foods.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in glucose concentrations measured by a glucose tolerance test. | 5 weeks

SECONDARY OUTCOMES:
Fetal growth | 5 weeks
  Measure abdominal circumference of fetus by ultrasound
Mean amplitude of glucose excursions | 5 weeks
  Measured with continuous glucose monitors

CONTACTS AND LOCATIONS:
Overall Officials: Paula Chandler-Laney, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No